CLINICAL TRIAL: NCT06559150
Title: A Phase II, Randomized, Double-Blind, Placebo- Controlled Study of Ensifentrine in Subjects With Non-Cystic Fibrosis Bronchiectasis
Brief Title: A Phase II Study of Ensifentrine in Non-Cystic Fibrosis Bronchiectasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RPL554-NCFB-220; 2024-514845-12 (EudraCT Number)
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Non-cystic Fibrosis Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1: Ensifentrine (Experimental)
  Interventions: Drug: Nebulized Ensifentrine Suspension; 3 mg
- Treatment Arm 2: Placebo (Placebo Comparator)
  Interventions: Drug: Nebulized Placebo Solution

INTERVENTIONS:
Drug: Nebulized Ensifentrine Suspension; 3 mg — Administered by a standard jet nebulizer, twice daily for a minimum of 24 weeks and up to a maximum of 156 weeks (3 years)
  Arms: Treatment Arm 1: Ensifentrine
Drug: Nebulized Placebo Solution — Administered by a standard jet nebulizer, twice daily for a minimum of 24 weeks and up to a maximum of 156 weeks (3 years)
  Arms: Treatment Arm 2: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study designed to assess the efficacy and safety of ensifentrine inhalation suspension (3 mg) delivered twice daily via standard jet nebulizer over at least 24 weeks, compared to placebo, in subjects with non-cystic fibrosis bronchiectasis (NCFBE).

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effect of ensifentrine vs placebo in addition to standard of care on pulmonary exacerbations, symptoms and quality of life in participants with NCFBE. The study is designed as a pulmonary exacerbation event-driven study where participants will be treated for ≥ 24 weeks and until at least 120 subjects have experienced at least 1 protocol-defined pulmonary exacerbation. Participants will be randomized to receive either ensifentrine suspension or placebo via standard jet nebulizer during the treatment period and neither participants nor study staff will know which a participant is receiving.

ELIGIBILITY:
Inclusion Criteria:

* Males are eligible to participate if they agree to use contraception as described in the contraceptive guidance from Screening and throughout the study and for at least 30 days after the last dose of blinded study medication
* Females are eligible to participate if they are not pregnant, not breastfeeding, and 1 of the following conditions apply:

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to follow the contraceptive guidance from Screening throughout the study and for at least 30 days after the last dose of blinded study medication
* Clinical history consistent with bronchiectasis (cough, chronic sputum production, and/or recurrent respiratory infections) confirmed by chest CT demonstrating bronchiectasis affecting 1 or more lobes. Confirmation may be based on prior chest CT within the prior 5 years; subjects whose past CT image records are not available will require chest CT scan during screening Notes: If a subject has no clinical history consistent with bronchiectasis, they may not be re-screened
* Current sputum producer with a history of chronic expectoration and able to provide sputum sample spontaneously at the clinic during screening
* ≥ 1 documented pulmonary exacerbation defined by an antibiotic prescription by a physician for the signs and symptoms of respiratory infections in the past 12 months before screening
* Capable of using the study nebulizer correctly
* Ability to perform acceptable spirometry in accordance with American Thoracic Society and European Respiratory Society guidelines

Exclusion Criteria:

* A diagnosis of COPD or a primary diagnosis of asthma, as judged by the investigator
* Bronchiectasis due to cystic fibrosis, hypogammaglobulinemia common variable immunodeficiency, severe immunodeficiency, or requirement for treatment with intravenous immunoglobulin
* Current smoker defined as by the Centers for Disease Control and Prevention (CDC)
* Former cigarette smokers with a history of cigarette smoking ≥ 10 pack years at Screening [number of pack years = (number of cigarettes per day / 20) × number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Pipe and/or cigar use cannot be used to calculate pack-year history. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Screening
* A diagnosis of primary ciliary dyskinesia
* Current treatment for nontuberculous mycobacterial lung infection, allergic bronchopulmonary aspergillosis, or tuberculosis
* Presence of acute exacerbation or acute infection that required acute treatment within 28 days of randomization
* Use of the following prohibited medications within the designated time periods:

  1. Immunomodulatory agents for any indication (including but not limited to the following: methotrexate, systemic corticosteroids, see adalimumab, azathioprine, dupilumab, cyclosporine) within 90 days prior to signing the ICF
  2. CFTR modulators (e.g., ivacaftor, lumacaftor, tezacaftor) within 1 week prior to signing the ICF
  3. Theophylline and PDE4 inhibitors (e.g., roflumilast, apremilast, crisaborole) within 48 hours prior to signing the ICF
  4. Brensocatib within 3 months or 5 half-lives, whichever is longer, prior to signing the ICF
  5. Ohtuvayre at any time prior to signing the ICF
* Initiated or altered therapy within 90 days of randomization with:

  1. oral or inhaled antibiotics as chronic treatment
  2. Cyclic antibiotics: defined as prescribed regular cycles of on antibiotic treatment and off antibiotic treatment (for example, but not limited to, 28 days on an antibiotic and 28 days off an antibiotic). Note: Subjects on cyclic antibiotics must be actively taking antibiotics for at least 7 days prior to randomization and through the day of randomization
* Initiated or altered therapy with ICS within 4 weeks prior to randomization
* Unable to withhold short-acting beta-agonists or short-acting muscarinic antagonists for ≥ 4 hours prior to spirometry
* Significant hemoptysis (≥ 300 mL or requiring blood transfusion) within 6 weeks prior to randomization
* Currently participating in or scheduled to participate in an intensive pulmonary rehabilitation program (a maintenance rehabilitation program is allowed if their schedule and procedure will be consistent for the duration of the study)
* Current or chronic history of unstable liver disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices or persistent jaundice, cirrhosis, or known hepatic or biliary abnormalities except for a diagnosis of Gilbert syndrome or asymptomatic gallstones Note: Chronic stable hepatitis B and C is not exclusionary if the subject otherwise meets study entry criteria
* History of or current malignancy of any organ system, treated or untreated within the past 5 years, except for localized basal or squamous cell carcinoma of the skin
* Estimated glomerular filtration rate (eGFR) < 30 mL/min
* Alanine aminotransferase (ALT) ≥ 2 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≥ 2 × ULN, alkaline phosphatase and/or bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN is acceptable only in subjects with a diagnosis of Gilbert's syndrome)
* Participation in any other interventional, clinical studies (drugs or devices) within 30 days before Day 1, or 5 half-lives, whichever is longer
* Intolerance of or hypersensitivity to ensifentrine or any of its excipients/components
* Current or history of drug or alcohol abuse within the past 5 years
* Significantly abnormal ECG finding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rate of protocol-defined pulmonary exacerbations (number of events per subject-year) | Through study completion (a maximum of 3 years from the date of randomization)

SECONDARY OUTCOMES:
Time to the onset of the first protocol-defined pulmonary exacerbation | Through study completion (a maximum of 3 years from the date of randomization)
Mean change from Baseline in Evaluating Respiratory Symptoms (E-RS) Cough and Sputum Domain score | Baseline, Week 6, Week 12, and Week 24
  The E-RS is a patient reported outcome that is derived from the EXAcerbation of Chronic Pulmonary Disease Tool (EXACT)-PRO in the participants e-diary, to quantify the severity of symptoms. The score ranges from 0 to 40 with a higher score representing more severe symptoms.
Mean change from Baseline in Saint George's Respiratory Questionnaire (SGRQ) score | Baseline, Week 6, Week 12, and Week 24
  SGRQ scores range from 0 to 100, with a higher score representing worse health.
Mean change from Baseline in quality of life - bronchiectasis questionnaire (QOL-B) Respiratory Symptoms Domain score | Baseline, Week 6, Week 12, and Week 24
  The QOL-B Respiratory Symptoms Domain score ranges from 0 to 100, with higher scores representing better functioning.
Mean change from Baseline in Chronic Airways Assessment Test (CAAT) score | Baseline, Week 6, Week 12, and Week 24
  CAAT scores range from 0-40 with a higher score representing worse health.
Mean change from Baseline in Percent of the predicted forced expiratory volume over 1 second (FEV1) | Baseline, Week 12, and Week 24
Incidence of Adverse Events | Through study completion (a maximum of 3 years from the date of randomization)
PK Sub-study only: Ensifentrine area under the curve from time 0 to 12 hours (AUC 0 -12) | Week 12, Week 18, and Week 24
PK Sub-study only: Ensifentrine maximum plasma drug concentration (Cmax) | Week 12, Week 18, and Week 24
Pharmacokinetic (PK) Sub-study only: Ensifentrine time to Cmax (tmax) post morning dose | Week 12, Week 18, and Week 24

CONTACTS AND LOCATIONS:
Locations (50):
- United States (28):
  - Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - So Cal Institute for Respiratory Diseases, Inc., Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - National Jewish Health Main Campus, Denver, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University at Saint Joseph Pulmonary Clinic, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - ASHA Clinical Research, Hammond, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center-Kansas City, Kansas City, Kansas
  - Massachusetts General Hospital- 55 Fruit St, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health Pulmonary and Critical Care Associates, P.C. - BRANY - PPDS, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Accellacare of Wilmington, Wilmington, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC) - PPDS, Charleston, South Carolina
  - Velocity Clinical Research - Spartanburg - PPDS, Spartanburg, South Carolina
  - Velocity Clinical Research - Union - PPDS, Union, South Carolina
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - The Respire Institute, Houston, Texas
  - UT Texas Health Science at Tyler, Tyler, Texas
  - TPMG Clinical Research, Williamsburg, Virginia
- Italy (5):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardi
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia
  - AOU Policlinico Gaspare Rodolico-San Marco Presidio Ospedaliero Gaspare Rodolico, Catania, Sicily
- Spain (8):
  - Hospital Universitario A Coruña, A Coruña, A Coruña
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
- United Kingdom (9):
  - Ninewells Hospital - PPDS, Dundee, Dundee
  - Queen Elizabeth University Hospital - PPDS, Glasgow, Glasgow
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - Queens Hospital Belfast, Belfast
  - Royal Papworth Hospital, Cambridge
  - Royal Infirmary of Edinburgh - PPDS, Edinburgh
  - Liverpool Heart and Chest Hospital - PPDS, Liverpool
  - Royal Brompton Hospital, London
  - Freeman Hospital, Newcastle-under-Lyme

IPD SHARING:
Plan to Share IPD: No